CLINICAL TRIAL: NCT02392546
Title: A Single Center, Placebo-controlled Trial to Evaluate the Effects of Elobixibat in Colonic Motor Functions in Patients With Chronic Idiopathic Constipation
Brief Title: Elobixibat Colonic Motor Function Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 000185
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — elobixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Elobixibat 10 mg (Experimental): elobixibat
  Interventions: Drug: elobixibat
- Elobixibat 15 mg (Experimental): elobixibat
  Interventions: Drug: elobixibat
- Elobixibat 20 mg (Experimental): elobixibat
  Interventions: Drug: elobixibat
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: elobixibat
  Arms: Elobixibat 10 mg; Elobixibat 15 mg; Elobixibat 20 mg
Drug: placebo
  Arms: Placebo

SUMMARY:
This is a randomized trial of 36 otherwise healthy patients with chronic idiopathic constipation. The purpose of the study is to compare the effects of daily single-dose oral elobixibat and placebo for 7 days on colonic motor effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-65 years of age
* Body Mass Index of 18-40 kg/m2
* Diagnosis of constipation for 12 or more weeks with symptom onset at least 6 months prior to the diagnosis and insufficient criteria to fulfill a diagnosis of irritable bowel syndrome (IBS), as defined by the Rome III criteria for Functional Constipation
* Stable concomitant medications defined as no changes in regimen for at least 2 weeks prior to the trial period

Exclusion Criteria:

* Structural or metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal (GI) disorders.
* Use of drugs or agents within the past 2 weeks that alter GI transit including laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, selective serotonin reuptake inhibitor and newer antidepressants
* Use of drugs or agents within the past 2 weeks that may add drowsiness and central nervous system (CNS) depression such as barbiturates, benzodiazepines, ethanol, lithium, opioids, buspirone, antihistamines, muscle relaxants, and other CNS depressants
* The patient has a history of bariatric surgery for treatment of obesity; surgery to remove a segment of the GI tract; or surgery of the abdomen, pelvic or retroperitoneal area during the 6 months prior to Screening; or appendectomy or cholecystectomy 3 months prior to screening; or other major surgery 1 month prior to Screening
* Clinical evidence (including physical exam) of clinically significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the trial. Any candidate participants with such disorder mentioned will be referred to their general physician
* The Hospital Anxiety and Depression Scale (HADS) will be used to exclude patients with significant affective disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Number of postprandial High Amplitude Propagated Contractions (HAPCs) | At Day 7
Postprandial Colonic Tone | At Day 7
Change in postprandial tone relative to fasting | At Day 7

SECONDARY OUTCOMES:
Fasting colonic tone | At Day 7
Colonic sensation threshold for first sensation | At Day 7
Colonic sensation threshold for gas | At Day 7
Colonic sensation threshold for pain | At Day 7
Total 48h fecal bile acid excretion | At Day 4-6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States